CLINICAL TRIAL: NCT00856960
Title: A Randomized, Double-Blind, Placebo-Controlled, 4-Treatment, 3-Period, Incomplete Block, Balanced Crossover Study to Evaluate the Effects of a Single Dose of Aliskiren and Losartan on Renal Blood Flow Measurements in Healthy Male Subjects
Brief Title: The Effect of Hypertension Medications on Renal Blood Flow Measurements in Healthy Males (MK-0000-127)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-127; 127; 2009_554
Record Dates: First submitted 2009-02-27; First posted 2009-03-06 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Aliskiren 600 mg
  Interventions: Drug: Aliskiren; Drug: Comparator: Placebo to Losartan
- 2 (Active Comparator): Aliskiren 150 mg
  Interventions: Drug: Aliskiren; Drug: Comparator: Placebo to Aliskiren; Drug: Comparator: Placebo to Losartan
- 3 (Active Comparator): Losartan 100 mg
  Interventions: Drug: Comparator: Losartan; Drug: Comparator: Placebo to Aliskiren
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo to Aliskiren; Drug: Comparator: Placebo to Losartan

INTERVENTIONS:
Drug: Aliskiren — Single dose of four 150 mg tablets (600 mg total) Aliskiren in one of three study periods. There will be at least 10 days between each study period.
  Arms: 1
Drug: Aliskiren — Single dose of one 150 mg tablet of Aliskiren in one of three study periods. There will be at least 10 days between each study period.
  Arms: 2
Drug: Comparator: Losartan — Single dose of one 100 mg tablet Losartan in one of three study periods. There will be at least 10 days between each study period.
  Arms: 3
Drug: Comparator: Placebo to Aliskiren — Three or four tablets placebo to Aliskiren 150 mg in one of three study periods. There will be at least 10 days between each study period.
  Arms: 2; 3; 4
Drug: Comparator: Placebo to Losartan — Single dose of placebo to Losartan 100 mg in one of three study periods. There will be at least 10 days between each study period.
  Arms: 1; 2; 4

SUMMARY:
This study will evaluate the effect of Aliskiren and Losartan on renal blood flow using PAH clearance, PC MRA and ASL MRI methodologies.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in generally good health
* Subject is willing to avoid unaccustomed strenuous exercise during the study
* Subject agrees to consume ONLY the study-specified diet during all domiciled periods
* Subject has been a non-smoker for at least 3 months prior to study
* Subject will refrain from smoking or using any tobacco products during the study
* Subject agrees to refrain from consuming alcohol or caffeine during the domiciled periods and agrees to limit alcohol and caffeine consumption throughout the study

Exclusion Criteria:

* Subject has contraindication to MRI scans
* Subject has a history of stroke, seizure, or major neurological disorders
* Subject uses illicit drugs or has a history of drug/alcohol abuse
* Subject has had major surgery, has donated or lost 1 unit of blood, or has been in another investigational study in the last 4 weeks
* Subject has a history of multiple and/or severe allergies to drugs or food

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
change in renal plasma flow as measured by PAH clearance and on renal blood flow as measured by ASL MRI after single-dose Aliskiren | 2-5 hours post dose of study drug

SECONDARY OUTCOMES:
change in renal plasma flow as measured by PAH clearance and on renal blood flow as measured by ASL MRI after single-dose Losartan | 2-5 hours post dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC